CLINICAL TRIAL: NCT01343927
Title: Yoga vs. Physical Therapy vs. Education for Chronic Low Back Pain in Minority Populations (Back to Health)
Brief Title: Yoga vs. Physical Therapy vs. Education for Chronic Low Back Pain in Minority Populations
Acronym: Back to Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-29779; R01AT005956 (NIH)
Record Dates: First submitted 2011-04-20; First posted 2011-04-28 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Chronic low back pain; Community health center; Yoga; Physical therapy; Minority populations; Health education
MeSH Terms: conditions — Health Education | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Yoga (Active Comparator): 12 weeks of weekly yoga classes plus 40 weeks of either drop-in classes or home practice.
  Interventions: Behavioral: Weekly yoga classes
- Physical Therapy (Active Comparator): 15 individual physical therapy treatment sessions over 12 weeks plus 40 weeks with either 5 booster sessions or home practice.
  Interventions: Behavioral: Individual physical therapy treatment
- Education (Active Comparator): "The Back Pain Helpbook" which gives exercises and tips for self-care pain management.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Weekly yoga classes — Manualized 12-week Hatha yoga intervention developed specifically for chronic low back pain in adult populations; classes meet once each week at community-based locations.
  Arms: Yoga
Behavioral: Individual physical therapy treatment — 12 weeks of fifteen individual physical therapy sessions divided as follows: Week 1 intake appointment; weeks 2-4 two appointments per week; weeks 5-12 one appointment per week.
  Arms: Physical Therapy
Behavioral: Education — Participants given "The Back Pain Helpbook" and periodic newsletters addressing back pain and self care.
  Arms: Education

SUMMARY:
A randomized controlled trial for chronic low back pain in predominantly minority populations with three treatment arms: yoga, physical therapy, and education. Four cohorts of participants will be randomized in a 2:2:1 ratio (yoga:physical therapy:education). Primary outcomes are pain intensity and measure of disability; secondary outcomes are pain medication use, treatment adherence, and health-related quality of life.

DETAILED DESCRIPTION:
Chronic low back pain (CLBP) affects 5-10% of U.S. adults annually and disproportionately impacts individuals from minority and low income backgrounds due to disparities in access and treatment. Our previous Yoga Dosing Study of 95 adults with chronic low back pain recruited from Boston Medical Center and affiliated community health centers showed that both once per week and twice per week yoga classes for 12 weeks were similarly effective for reducing pain and improving back related function. We concluded that due to the superior convenience and lower cost of once per week compared to twice per week classes, a once per week yoga protocol was optimal for the current study. Evidence from multiple studies supports a moderate benefit in CLBP for exercise therapy individually-delivered by a physical therapist. Moreover, physical therapy is the most common, reimbursed, non-pharmacologic treatment recommended by physicians for CLBP. However, no studies to date have done a head-to-head comparison of the effectiveness of yoga and physical therapy for CLBP. To ultimately reduce disparities in CLBP for minority populations, patients, providers, and health insurers need to know how a complementary therapy such as yoga compares in effectiveness to more well established treatments such as physical therapy (PT) and education. If yoga is superior to education and has similar effectiveness as PT but costs less with greater adherence, the potential therapeutic and economic implications would be substantial. Alternatively, if yoga is inferior, this information will help guide better treatment decisions and reduce unnecessary expenditures on inferior treatments.

The present study (Back to Health) is a 52 week comparative effectiveness randomized controlled trial of once per week yoga classes, individually delivered physical therapy (PT), and education for chronic low back pain (CLBP) in 320 individuals from predominantly minority backgrounds recruited from Boston Medical Center and affiliated community health centers. The 52 week trial starts with an initial 12 week Treatment Phase followed by a 40 week Maintenance Phase. Back to Health has the following three specific aims:

1. In the 12 week Treatment Phase, we will enroll 320 adults with chronic low back pain(CLBP) from predominately low-income minority communities and compare the effectiveness (co-primary endpoints pain and function) between (1) a standardized protocol of one yoga class per week; (2) a standardized exercise therapy protocol based on an evidence-based clinical guidelines individually delivered by a physical therapist; and (3) an educational book on self-care for CLBP
2. For adults with CLBP who have completed the initial 12 week yoga or physical therapy(PT) Treatment Phases, compare effectiveness (co-primary endpoints pain and function)between patients participating in a structured yoga maintenance program, a structured PT maintenance program, or no structured maintenance program.
3. Determine the cost-effectiveness of yoga, PT, and education for adults with CLBP at 12 weeks, 6 months, 9 months, and one year from three perspectives: society, third party payers, and the participant.

For the 12 week Treatment Phase, participants are randomized in a 2:2:1 ratio into (1) a standardized once per week hatha yoga class supplemented by home practice; (2) a standardized evidence-based exercise therapy protocol individually delivered by a physical therapist and supplemented by home practice; and (3) education delivered through a self-care book. The study co-primary endpoints are mean pain intensity over the previous week measured on a 11 point numerical rating scale and back-specific function measured using the 23 point modified Roland Morris Disability Questionnaire. We hypothesize: (1) yoga will be noninferior to physical therapy; and (2) both yoga and physical therapy will be superior to education.

For the 40 week Maintenance Phase, yoga participants will be re-randomized in a 1:1 ratio to either a structured ongoing maintenance yoga program or no maintenance yoga program. Similarly, physical therapy participants will be re-randomized in a 1:1 ratio to either a structured ongoing maintenance PT program or no maintenance PT program. Education participants will be encouraged to continue to review and follow the recommendations of their educational materials. We hypothesize: (1) maintenance yoga will be non-inferior to maintenance PT; (2) maintenance yoga and maintenance PT will be superior to no yoga maintenance and no PT maintenance, respectively; and (3) maintenance yoga and maintenance PT will both be superior to education.

We will also take advantage of a comprehensive integrated set of patient databases, self-report cost data, and study records to compare at 3 months, 6 months, 9 months, and one year the cost-effectiveness of yoga, physical therapy, and education from three perspectives: society,third-party payer, and the participant. Qualitative data from interviews and focus groups will add subjective detail to complement quantitative data.

Results from the Back to Health Study will help determine whether it is justifiable for yoga, currently a "complementary" therapy, to become an acceptable "mainstream" treatment for chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Current non-specific low back pain persisting for at least 12 weeks
* 18-64 years old
* Mean low back pain intensity for the previous week of 4 or greater on a 0 to 10 numerical rating scale (0=no pain to 10=worst possible pain)
* English fluency sufficient to follow treatment instructions and answer survey questions.

Exclusion Criteria:

* New CLBP treatments started within the previous month or anticipated to begin in the next 3 months
* Known pregnancy
* Inability to understand English at a level necessary to understand treatment instructions and survey questions
* Previous back surgery or back fracture
* Specific CLBP pathologies (including spinal canal stenosis, severe scoliosis, spondylolisthesis, ankylosing spondylitis, large herniated disk)
* Severe or progressive neurological deficits
* Sciatica pain equal to or greater than back pain
* Active or recent cervical radiculopathy
* Active or planned worker's compensation, disability, or personal injury claims
* Lack of consent
* Significant participation in yoga or physical therapy in the last six months
* Has read The Back Pain Helpbook or the Back Book in the previous six months
* The principal investigator judges the participant to be unable to participate in the study due to serious medical and/or psychiatric comorbidities
* Has previously participated in the Yoga Dosing Study or the Physical Therapy Pilot
* Plans to move out of the Boston area in the next year

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Average Pain intensity in previous week | 12 wks
  Intensity of pain in previous week as measured on a 10 point numerical scale (0-10).
Change from Baseline in Modified Roland Morris questionnaire for Back pain specific disability | 12 wks
  Utilize modified 23-point scale standardized Roland Morris questionnaire to asses back pain specific disability.

SECONDARY OUTCOMES:
Change from baseline in Pain Medication use in the previous week | 12wks
  Specific self-reported pain medication use in previous week.
Satisfaction with assigned intervention at 12 weeks | 12 wks
  Self-reported satisfaction with intervention using 5-point Likert scale from very dissatisfied to very satisfied
Global improvement in back pain at 12 weeks | 12wks
  Self-reported rating of global improvement since start of study using 7-point Likert scale from extremely worsened to extremely improved
Change from Baseline for Health related Quality of Life using SF-36 survey | 12wks
  Use standardized Quality of life SF-36 questionnaire.
Work productivity | 12wks
  Use standardized Work Productivity and Activity Impairment questionnaire to assess employment status and productivity

OTHER OUTCOMES:
Number of participants with Adverse Events as a measure of safety and treatment adherence | 12wks
  Identify and assess self reported and unanticipated adverse events over the course of the study as a measure of safety and treatment adherence.
Treatment adherence (class/session attendance) | 12wks
  Assess treatment adherence according to attendance during 12 week intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Saper, MD, MPH, Principal Investigator — Boston University School of Medicine/ Boston Medical Center
Locations (8):
- United States (8):
  - Boston Medical Center, Boston, Massachusetts
  - South End Community Health Center, Boston, Massachusetts
  - Dimock Health Center, Boston, Massachusetts
  - Dorchester House MultiService Center, Dorchester, Massachusetts
  - Codman Square Health Center, Dorchester, Massachusetts
  - Upham's Corner Health Center, Dorchester, Massachusetts
  - Greater Roslindale Medical and Dental Center, Roslindale, Massachusetts
  - South Boston Community Health Center, South Boston, Massachusetts

REFERENCES:
- [Background] Saper RB, Sherman KJ, Cullum-Dugan D, Davis RB, Phillips RS, Culpepper L. Yoga for chronic low back pain in a predominantly minority population: a pilot randomized controlled trial. Altern Ther Health Med. 2009 Nov-Dec;15(6):18-27. PMID 19943573
- [Background] Saper RB, Boah AR, Keosaian J, Cerrada C, Weinberg J, Sherman KJ. Comparing Once- versus Twice-Weekly Yoga Classes for Chronic Low Back Pain in Predominantly Low Income Minorities: A Randomized Dosing Trial. Evid Based Complement Alternat Med. 2013;2013:658030. doi: 10.1155/2013/658030. Epub 2013 Jun 26. PMID 23878604
- [Derived] Joyce C, Kelly KC, Gurnani S, Sherman KJ, Roseen EJ, Saper RB. "In Class We Were All One." A Qualitative Exploration of Yoga and Educational Interventions for Predominantly Low-Income and Minority Adults with Chronic Low Back Pain. J Integr Complement Med. 2022 Nov;28(11):870-877. doi: 10.1089/jicm.2022.0557. Epub 2022 Aug 1. PMID 35914101
- [Derived] Joyce CT, Chernofsky A, Lodi S, Sherman KJ, Saper RB, Roseen EJ. Do Physical Therapy and Yoga Improve Pain and Disability through Psychological Mechanisms? A Causal Mediation Analysis of Adults with Chronic Low Back Pain. J Orthop Sports Phys Ther. 2022 Jul;52(7):470-483. doi: 10.2519/jospt.2022.10813. Epub 2022 May 18. PMID 35584010
- [Derived] Marshall A, Joyce CT, Tseng B, Gerlovin H, Yeh GY, Sherman KJ, Saper RB, Roseen EJ. Changes in Pain Self-Efficacy, Coping Skills, and Fear-Avoidance Beliefs in a Randomized Controlled Trial of Yoga, Physical Therapy, and Education for Chronic Low Back Pain. Pain Med. 2022 Apr 8;23(4):834-843. doi: 10.1093/pm/pnab318. PMID 34698869
- [Derived] Joyce C, Roseen EJ, Keysor JJ, Gross KD, Culpepper L, Saper RB. Can Yoga or Physical Therapy for Chronic Low Back Pain Improve Depression and Anxiety Among Adults From a Racially Diverse, Low-Income Community? A Secondary Analysis of a Randomized Controlled Trial. Arch Phys Med Rehabil. 2021 Jun;102(6):1049-1058. doi: 10.1016/j.apmr.2021.01.072. Epub 2021 Feb 5. PMID 33556352
- [Derived] Roseen EJ, Gerlovin H, Felson DT, Delitto A, Sherman KJ, Saper RB. Which Chronic Low Back Pain Patients Respond Favorably to Yoga, Physical Therapy, and a Self-care Book? Responder Analyses from a Randomized Controlled Trial. Pain Med. 2021 Feb 4;22(1):165-180. doi: 10.1093/pm/pnaa153. PMID 32662833
- [Derived] Berlowitz J, Hall DL, Joyce C, Fredman L, Sherman KJ, Saper RB, Roseen EJ. Changes in Perceived Stress After Yoga, Physical Therapy, and Education Interventions for Chronic Low Back Pain: A Secondary Analysis of a Randomized Controlled Trial. Pain Med. 2020 Oct 1;21(10):2529-2537. doi: 10.1093/pm/pnaa150. PMID 32500130
- [Derived] Roseen EJ, Gerlovin H, Femia A, Cho J, Bertisch S, Redline S, Sherman KJ, Saper R. Yoga, Physical Therapy, and Back Pain Education for Sleep Quality in Low-Income Racially Diverse Adults with Chronic Low Back Pain: a Secondary Analysis of a Randomized Controlled Trial. J Gen Intern Med. 2020 Jan;35(1):167-176. doi: 10.1007/s11606-019-05329-4. Epub 2019 Oct 30. PMID 31667747
- [Derived] Saper RB, Lemaster C, Delitto A, Sherman KJ, Herman PM, Sadikova E, Stevans J, Keosaian JE, Cerrada CJ, Femia AL, Roseen EJ, Gardiner P, Gergen Barnett K, Faulkner C, Weinberg J. Yoga, Physical Therapy, or Education for Chronic Low Back Pain: A Randomized Noninferiority Trial. Ann Intern Med. 2017 Jul 18;167(2):85-94. doi: 10.7326/M16-2579. Epub 2017 Jun 20. PMID 28631003
- [Derived] Saper RB, Sherman KJ, Delitto A, Herman PM, Stevans J, Paris R, Keosaian JE, Cerrada CJ, Lemaster CM, Faulkner C, Breuer M, Weinberg J. Yoga vs. physical therapy vs. education for chronic low back pain in predominantly minority populations: study protocol for a randomized controlled trial. Trials. 2014 Feb 26;15:67. doi: 10.1186/1745-6215-15-67. PMID 24568299